CLINICAL TRIAL: NCT03101423
Title: Monitoring of Chimerism After Transplantation in Patients With β Thalassemia Major and the Treatment Strategies for the Reduction of Chimerism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Liang Bo, Principal Investigator, First Affiliated Hospital of Guangxi Medical University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LBo
Record Dates: First submitted 2017-03-26; First posted 2017-04-05 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Beta Thalassemia Major
Keywords: thalassemia; transplantation; chimerism; donor ymphocytes
MeSH Terms: conditions — beta-Thalassemia; Thalassemia | interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interleukin-2 (Active Comparator): interleukin-2 treatment per month
  Interventions: Drug: Interleukin-2
- DLI (Active Comparator): donor lymphocyte infusion (DLI) treatment per month
  Interventions: Drug: Donor Regulatory T-Lymphocytes

INTERVENTIONS:
Drug: Interleukin-2 — On +60 day after transplantation,check patients with STR more than or equal to 90%. transplantat interleukin-2 treatment per month
  Arms: interleukin-2
Drug: Donor Regulatory T-Lymphocytes — On +60 day after transplantation,check patients with STR less than 90%. Donor Regulatory T-Lymphocytes infusion (DLI) treatment per month
  Arms: DLI

SUMMARY:
Hematopoietic stem cell transplantation is currently the only way to cure thalassemia, one of its main obstacles is the rejection after transplantation, chimerism continued to decline, which eventually lead to transplant failure. chimerism is a key indicator of the succession of immune response, which is a key indicator for predicting the failure of hematopoietic stem cell transplantation and provides an important basis for early detection of rejection. Transplantation of continuous chimerism can detect early unstable chimeras and rejection.The chimerism rates after transplantation were continuously monitored using fluorescence labeled multiplex PCR amplification of short tandem repeats (STR-PCR)

,and then follow our STR different rates for early interventional therapy to prevent further reduction in chimerism leading to lead to graft failure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of thalassemia major
2. There is no restriction on age or gender.
3. Underwent allogeneic hematopoietic stem cell transplantation, including sibling transplantation, unrelated transplantation and haploidentical transplantation.
4. On +45 day after transplantation, check patients with STR less than 80%.
5. Patients underwent reduce of dosage with a failure treatment by
6. Body condition score (ECOG score) is less than or equal to 1 point who meet follow-up conditions.

Exclusion Criteria:

Complicated with severe cardiac insufficiency and cardiac ejection fraction (EF) was lower than 50%. Complicated with severe pulmonary insufficiency (obstructive and / or restrictive ventilatory disorders). Complicated with severe liver function damage and liver function index (ALT or TBIL) is more than 2 times of the upper limit of the normal value. Complicated with severe renal dysfunction and renal function index (Cr or BUN) is 2 times of the upper limit of the normal value. Complicated with severe active bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Chimerism after transplantation were monitored using fluorescence labeled multiplex PCR amplification of short tandem repeats (STR-PCR) | Change from chimerism rate at 2-3 months after different treatment
  β thalassemia major patients underwent reduced chimerism rate after allogeneic hematopoietic stem cell transplantation were collected and the chimerism rates after transplantation were continuously monitored using fluorescence labeled multiplex PCR amplification of short tandem repeats (STR-PCR).Monitoring once every 20-30 days after allogeneic hematopoietic stem cell transplantation.For patients with reduced chimerism, the results were grouped.We monitor STR-PCR once every 20-30 days after different treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China